CLINICAL TRIAL: NCT07061288
Title: An Open-label, Phase 1, Single Ascending Dose-Finding Study to Characterize the Safety, Tolerability, and Pharmacokinetics of a Long Acting Injectable KarXT Formulation in Participants With Schizophrenia
Brief Title: A Study to Evaluate the Dose Levels, Safety, and Drug Levels of Single KarXT Intramuscular Injection in Participants With Schizophrenia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0016
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: KarXT; Long-acting injectable (LAI); Cobenfy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of KarXT (Experimental)
  Interventions: Drug: KarXT

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510

SUMMARY:
The purpose of this study is to evaluate the dose levels, safety, and drug levels of KarXT intramuscular injection in participants with Schizophrenia

ELIGIBILITY:
Inclusion Criteria

* Participants must have a primary diagnosis of schizophrenia, as confirmed by psychiatric evaluation based on Diagnostic and Statistical Manual of Mental Disorders (5th Edition, Text Revision) (DSM-5-TR) criteria and Mini International Neuropsychiatric Interview (MINI) (version 7.0.2).
* Participants must have a Positive and Negative Syndrome Scale (PANSS) total score ≤ 80 and a Clinical Global Impression - Severity (CGI-S) score ≤ 4 at both screening and baseline.
* Participants must have a body mass index (BMI) between 18 and 40 kg/m².
* Participants should be willing and able, as determined by the investigator, to discontinue all antipsychotic medications prior to the baseline visit and must be able to comply with all protocol requirements.

Exclusion Criteria

* Participants must not have newly diagnosed schizophrenia or a first treated episode of schizophrenia.
* Participants must not have any other DSM-5-TR disorder diagnosed within the past 12 months, such as major depressive disorder or bipolar disorder.
* Participants must not have a history of alcohol or drug use disorder within the past 12 months or those with clinically significant disease or disorder that would jeopardize their safety or affect the validity of study results.
* Participants must not be at risk for suicidal behavior.
* Female participants must not be pregnant or breastfeeding.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-06-21 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 3 weeks
Number of participants with adverse events of special interest (AESIs) | Up to 3 weeks
Number of participants with serious adverse events (SAEs) | Up to 3 weeks

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Up to 15 weeks
Time to maximum concentration (Tmax) | Up to 15 weeks
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) | Up to 15 weeks
Area under the plasma concentration-time curve from time zero to infinity (AUC(INF)) | Up to 15 weeks
Area under the plasma concentration-time curve from time zero to 672 hours (AUC(0-672)) | Up to 15 weeks
Apparent terminal phase half-life (T-HALF) | Up to 15 weeks
Apparent total body clearance (CLT/F) | Up to 15 weeks
Apparent volume of distribution of terminal phase (Vz/F) | Up to 15 weeks
Number of participants with AEs | Up to 3 weeks
Number of participants with AESIs | Up to 3 weeks
Number of participants with SAEs | Up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (8):
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Hassman Research Institute Marlton Site, Marlton, New Jersey
  - Community Clinical Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07061288.html